CLINICAL TRIAL: NCT02190981
Title: Point of Care Ultrasound for Suspected Small Bowel Obstruction in the Emergency Department
Status: Completed | Type: Observational
Sponsor: WellSpan Health (Other)
Collaborators: University of California, Irvine (Other); Christiana Care Health Services (Other)
Responsible Party: Principal Investigator, Brent Becker, Emergency Physician - Wellspan Health York Hospital, WellSpan Health
Other Study IDs: 615362-1
Record Dates: First submitted 2014-07-10; First posted 2014-07-15 (Estimated); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Small Bowel Obstruction
Keywords: Small bowel obstruction; Ultrasound; Emergency department
MeSH Terms: conditions — Emergencies | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ultrasound for Small Bowel Obstruction: Emergency department patients undergoing point-of-care ultrasound to evaluate for suspected small bowel obstruction
  Interventions: Device: Ultrasound for Small Bowel Obstruction

INTERVENTIONS:
Device: Ultrasound for Small Bowel Obstruction — Point-of-care ultrasound to evaluate emergency department patients for suspected small bowel obstruction

SUMMARY:
The primary purpose of this study is to determine the accuracy of ultrasound in diagnosing small bowel obstruction in emergency department patients, as compared to the criterion standards of computed tomography, operative reports, or discharge diagnosis.

The secondary purposes of the study include evaluation of the effect of ultrasound for small bowel obstruction on the patient length of stay in the emergency department and the diagnostic utility of specific ultrasound findings in the diagnosis of small bowel obstruction. The study will also examine the inter-rater agreement between point-of-care sonographers' interpretation and blinded reviewers' interpretation of the ultrasound images.

DETAILED DESCRIPTION:
Background:

An estimated 15% of emergency department (ED) patients admitted to a surgical unit with abdominal pain are ultimately diagnosed with small bowel obstruction (SBO) (1). The work up of patients with possible SBO is directed by the patient history, physical examination and pre-test probability. Relatively insensitive abdominal x-rays (AXR) are commonly ordered as a screening test, but computed tomography (CT) imaging is often necessary to confirm or exclude the diagnosis of SBO. This diagnostic process is time consuming, costly and exposes the patient to ionizing radiation.

Interest in point-of-care (POC) ultrasonography (US) for the evaluation of suspected SBO has increased in recent years. A growing body of literature suggests US is more sensitive and specific compared to AXR in the diagnosis of SBO (1-3). US also confers the benefits of less radiation exposure and more rapid decision-making. CT is generally considered the diagnostic criterion standard for SBO, but effective use of POC US may reduce the need for CT imaging and expedite the care of patients with suspected SBO.

Currently, there are five emergency physicians (EP) on staff in the York Hospital ED who are fellowship trained in POC US. These physicians are fully credentialed and are already performing ED based evaluations for small bowel obstruction. We intend to evaluate the performance of EP-performed POC US in the diagnosis of SBO in ED patients. This study would primarily investigate the accuracy of ultrasound as compared to the criterion standard of abdominal CT results, intraoperative diagnosis, or discharge diagnosis.

Study design:

This will be a prospective, observational study of adult ED patients suspected of having a SBO. ED nurses, residents, and attendings will perform the initial screening for potential enrollees. Once consented and enrolled, a study sonographer will interview and examine the patient, preferably before labs and AXR results. The ultrasound must be completed and adequate images obtained before advanced imaging modalities are completed. Ultrasound of all four abdominal quadrants will be performed using the "mowing the lawn" technique described previously in the literature (4).

The ultrasounds will be performed by all five of the US fellowship-trained EPs on staff, as well as two current emergency ultrasound fellows and three emergency medicine residents. All will participate in the identification, consent, and enrollment of patients in the study.

Trainees will undergo an hour-long educational session on POC US for SBO involving both lectures and hands on training. Methods for proper consent and data collection will be included. Blinded review of each ultrasound is already planned as a component of the study design and treatment decisions will not be made based on trainees ultrasounds unless supervised by a credentialed faculty member. The five faculty EP sonographers are already fully credentialed in POC ultrasound and familiar with the technique for SBO. No additional ultrasound training will be required for these participants.

A "Bedside" standardized data collection form will be used at the bedside to record ultrasound findings and clinical information. The sonographer will designate the ultrasound as "positive for small bowel obstruction," "negative for small bowel obstruction," or "indeterminate" based on the exam and ultrasound findings.

A second sonographer, blinded to all clinical information and the primary sonographer's ultrasound interpretation, will review the de-identified ultrasound images remotely. This over-reading sonographer will record his interpretation and secondary findings on a "Blinded Reviewer" standardized data collection sheet. Only fully credentialed, fellowship-trained EPs will serve as secondary, blinded reviewers. Current fellows and residents involved in the study will not review ultrasound images in this capacity.

CT imaging, intraoperative reports, and discharge diagnosis will be utilized to determine final outcome of patient's clinical course. At this time, a third "Follow Up" standardized data collection sheet will be used to record patient outcomes and demographic information.

In general, CT reports will be used as the criterion standard to which POC US findings will be compared and by which sensitivity/specificity will be calculated. If no CT is obtained, then operative report(s) will serve as the criterion standard. If the patient does not receive CT imaging or undergo surgical intervention, then the discharge diagnosis will serve as the criterion standard.

Study population and recruitment methods:

The study population will include adult patients presenting to the emergency department with abdominal pain and a clinical suspicion of SBO. A treating attending physician or resident will evaluate the patient. If there is a concern for SBO, the treating physician will contact one of the ultrasound credentialed EP sonographers to perform a POC US to evaluate for possible SBO. This process is the current practice standard in the ED.

At this point, the EP sonographer will approach the patient regarding the study. If the patient agrees to participate, the EP sonographer will obtain informed consent. Of note, the patient's treatment is unchanged, regardless of whether or not he/she consents to participation in the study. The POC US will be obtained in either case, as this is standard clinical practice in the ED. Agreeing to participate will simply allow the study team to collect data and review their chart upon discharge from the hospital. The study sonographer will obtain consent.

Data to be collected:

The following data will be recorded:

* Patients initials
* Patient Medical Record Number (MRN)/Financial Number (FIN)
* Age
* Sex
* Height
* Weight
* Chief complaint
* Presence/location of abdominal pain
* Symptom duration
* Associated symptoms (i.e. nausea/vomiting, diarrhea, etc.)
* Visualization of the small bowel?
* Maximum inner diameter of the small bowel?
* Presence of "to-and-fro" peristalsis?
* Edema of the wall of the small bowel?
* Presence of free fluid surrounding the small bowel?
* Presence of sonographic transition point?
* Diagnostic impression of the sonographer
* Diagnostic impression of the blinded reviewer
* XR findings
* CT diagnosis
* Operative report classification
* Time of patient placement in ED bed
* Time of consultation or ED discharge
* Discharge diagnosis

Data analysis:

For the primary outcome, data will be used to calculate the sensitivity and specificity of POC US for the diagnosis of SBO compared to the criterion standard of CT or operative report.

For secondary outcomes, likelihood ratios for specific ultrasound findings will be determined. Inter-rater agreement between the bedside sonographer and the blinded reviewer will be calculated using Cohen's kappa coefficient. Continuous, time-to-disposition data will be compared utilizing a two-tailed t-test.

Statistical analysis will be performed using SPSS software (IBM, Armonk, NY).

Risks and risk management:

There are minimal risks to patients participating in this study since ultrasound is non-invasive and known to be safe. There is a slight risk of the participants' privacy or confidentiality being breached. Standard precautions will be taken to ensure privacy and confidentiality is maintained during the study.

Benefits:

Patients whose ultrasound is highly suspicious for small bowel obstruction may be referred directly to surgery without further imaging being performed. In these instances study patients would benefit from reduced radiation exposure and faster referral for appropriate surgical care. The results of this study may be used to improve future patient care.

Compensation / incentives and research-related costs:

No compensation will be given to the participants. There will be no research-related costs.

Alternative procedures:

Patients who refuse to participate in the study will not have the quality of their treatment affected in any way.

Research materials, records, and confidentiality:

Research records will be stored in locked offices, filing cabinets, and computers using password-protected encryption.

Subject informed consent:

We will seek documented informed consent and Heath Insurance Portability and Accountability Act (HIPAA). ED patients meeting all of the inclusion and exclusion criteria will be asked if they would like to participate in the study by a research sonographer at the time of the ultrasound.

If the patient agrees to participate, the informed consent document will be given to them for their review. If patient declines to participate they will continue their treatment course in the Emergency Department.

References of relevant literature:

1. Taylor, Mark R. and Nadim Lalani. Adult Small Bowel Obstruction. Academic Emergency Medicine. 2013; 20:528-544.
2. Jang, Timothy B, et al. Bedside Ultrasonography for the Detection of Small Bowel Obstruction in the Emergency Department. Journal of Emergency Medicine. 2011;28:676-678.
3. Suri, S, et al. Comparative evaluation of plain films, ultrasound, and CT in the diagnosis of intestinal obstruction. Acta Radiologica. 40(1999): 422-428.
4. Mallin, Mike and Matthew Dawson. Introduction to Bedside Ultrasound: Volume 2. Emergency Ultrasound Solutions. 20 May 2013.
5. Ko, Tae, et al. Small Bowel Obstruction: Sonographic Evaluation. Radiology. 1993;188:649-653.
6. Ogata, Masaaki, James R. Mateer, and Robert E. Condon. Prospective Evaluation of Abdominal Sonography for the Diagnosis of Bowel Obstruction. Annals of Surgery. 1996;223(3):237-241.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or greater
* Abdominal pain with clinical suspicion for small bowel obstruction

Exclusion Criteria:

* Less than 18 years of age
* Lack of decision-making capacity or cannot provide consent
* Pregnancy
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult emergency department patients at a university-affiliated, community teaching hospital with suspected small bowel obstruction
Sampling Method: Non-Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Diagnostic Accuracy of Point-of-care Ultrasound for Small Bowel Obstruction | 2 years
  The performance of point-of-care ultrasound for small bowel obstruction will be evaluated by comparing each ultrasound to the criterion standard of computed tomography (CT) for each enrolled patient. If a CT is not obtained, then operative report/findings or discharge diagnosis will be used as the criterion standard to which the ultrasound will be compared.
  Using the criterion standard as the definitive diagnosis for each patient (i.e. presence or absence of small bowel obstruction), each ultrasound will be classified as a true positive, true negative, false positive or false negative. This data will be used to calculated the sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV) and accuracy of point-of-care ultrasound for the diagnosis of small bowel obstruction.

SECONDARY OUTCOMES:
Incidence/Likelihood Ratios of Specific Sonographic Findings of Small Bowel Obstruction | 2 years
  Specific sonographic findings include:
  * Small bowel diameter >25 mm
  * "To-and-Fro" peristalsis
  * Small bowel wall edema
  * Presence of intrabdominal free fluid
  * Presence of sonographic transition point (defined as the location between dilated small bowel proximal to the obstruction and decompressed small bowel distal to the obstruction)
Inter-rater Agreement | 2 years
  The study will quantify the rate of inter-rater agreement between the clinician performing the point-of-care ultrasound and a blinded reviewer of the ultrasound images.
Patient Length of Stay/Time to Disposition | 2 years
  The study will measure the time to disposition of ED patients undergoing a point of care ultrasound for small bowel obstruction and determine how the ultrasound effects time to patient disposition.

CONTACTS AND LOCATIONS:
Overall Officials: Brent A Becker, MD, Principal Investigator — Wellspan Health York Hospital
Locations (3):
- United States (3):
  - University of California Irvine Medical Center, Orange, California
  - Christana Hospital, Wilmington, Delaware
  - Wellspan Health York Hospital, York, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Taylor MR, Lalani N. Adult small bowel obstruction. Acad Emerg Med. 2013 Jun;20(6):528-44. doi: 10.1111/acem.12150. PMID 23758299
- [Background] Jang TB, Schindler D, Kaji AH. Bedside ultrasonography for the detection of small bowel obstruction in the emergency department. Emerg Med J. 2011 Aug;28(8):676-8. doi: 10.1136/emj.2010.095729. Epub 2010 Aug 22. PMID 20732861
- [Background] Suri S, Gupta S, Sudhakar PJ, Venkataramu NK, Sood B, Wig JD. Comparative evaluation of plain films, ultrasound and CT in the diagnosis of intestinal obstruction. Acta Radiol. 1999 Jul;40(4):422-8. doi: 10.3109/02841859909177758. PMID 10394872
- [Background] Ko YT, Lim JH, Lee DH, Lee HW, Lim JW. Small bowel obstruction: sonographic evaluation. Radiology. 1993 Sep;188(3):649-53. doi: 10.1148/radiology.188.3.8351327.
- [Background] Ogata M, Mateer JR, Condon RE. Prospective evaluation of abdominal sonography for the diagnosis of bowel obstruction. Ann Surg. 1996 Mar;223(3):237-41. doi: 10.1097/00000658-199603000-00002. PMID 8604902
- [Derived] Becker BA, Lahham S, Gonzales MA, Nomura JT, Bui MK, Truong TA, Stahlman BA, Fox JC, Kehrl T. A Prospective, Multicenter Evaluation of Point-of-care Ultrasound for Small-bowel Obstruction in the Emergency Department. Acad Emerg Med. 2019 Aug;26(8):921-930. doi: 10.1111/acem.13713. Epub 2019 Mar 12. PMID 30762916